CLINICAL TRIAL: NCT06602986
Title: Measuring the Density of Iodine in Lipiodol Depositions: Detecting an Invisible Residual Tumor After Conventional Transarterial Chemoembolization for Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, DR.Talha Arshad, Professor Radiology, Pak Emirates Military Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: PakEmirates AFIRI
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- International study (Experimental): Hepatocellular carcinoma (HCC) is associated with considerable morbidity and mortality with a high prevalence in developing countries including Pakistan1. Statistics from Pakistan indicate that the cancer is among the top five causes of cancer deaths nationally and the commonest cancer in adult males with respect to frequency of diagnosis2. Risk factors implicated in our population are chronic hepatitis B and C infection, alcohol consumption, autoimmune hepatitis, Wilson disease and alpha-1 anti-trypsin deficiency as the commonest causes3. It is projected that lifestyle modifications including eating habits and increase in the frequency of hepatitis B and C infections would increase the incidence of the disease by threefold in the next decade4.
  The treatment options for the disease are diverse depending on the tumor size, location, time of diagnosis and associated co-morbidities. Small tumor with local restriction are offered surgical options including resection and/or tr
  Interventions: Diagnostic Test: TACE

INTERVENTIONS:
Diagnostic Test: TACE — study was carried out in our setup for two major reasons. One was to decrease reliance on DSA since it is a costly investigation in our medical setups and the facility is not available except for a few centers of excellence which creates issues with treatments plan of patients admitted for treatment using TACE and subsequent follow-up visits to assess the presence or absence of HCC tumors. The mean age of patients in our treatment group was in the early sixties. This is in line with the median age of diagnosis for HCC globally as evidenced by studies done by Mc Glynn et al12 and Konyn et al13. Gender distribution was predominantly male in our study group in line with available literature14. The Child Pugh classification which quantifies severity of chronic liver disease by assessing clinical parameters was used in our study as well15. Since the inclusion criteria and procedural requirement required normal bilirubin levels, all subjects in the study protocol were in Class A16.
  The prima

SUMMARY:
ABSTRACT Objective: To detect presence of a residual tumor in patients of hepatocellular carcinoma (HCC) treated with Lipiodol based conventional trans arterial chemoembolization (cTACE) using density measurements on follow-up computed tomography (CT) scans Study Design: Prospective observational interventional study Place and Duration of Study: Interventional Radiology department of Armed Forces Institute of Radiology and Imaging (AFIRI) from April 2023-March 2024 Methodology: 96 patients undergoing conventional TACE were included in the study and followed up for residual tumor or tumor free status assessment using density measurement for iodine depositions using CT scan analysis and compared with gold standard digital subtraction angiography (DSA). Primary variables measured were comparison of enhancement scores between those with a residual tumor versus tumor free as well as the volume of iodine depositions in the arterial and venous phase between both groups. Sensitivity and specificity of the CT scan in assessing tumor diagnosis was compared with the gold standard digital subtraction angiography.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HCC disease
* Must be able to swallow tablets

Exclusion Criteria:

* Insulin dependent diabetes
* Thyroid disease

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-10-12 (Estimated); Primary Completion 2025-02-12 (Estimated); Study Completion 2025-07-13 (Estimated)

PRIMARY OUTCOMES:
Measuring the density of Iodine in Lipiodol depositions: Detecting an Invisible Residual Tumor after Conventional Transarterial Chemoembolization for Hepatocellular carcinoma | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- PakEmiratesMH, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No